CLINICAL TRIAL: NCT03956797
Title: Long Term Evaluation of the Safety and Efficacy of Cooling Anesthesia for Local Anesthesia During Intravitreal Injection (COOL-2)
Brief Title: Long Term Safety of Cooling Anesthesia for Intravitreal Injection
Acronym: COOL-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recens Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: COOL-2.0
Record Dates: First submitted 2019-04-25; First posted 2019-05-21 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Anesthesia, Local; Intravitreal Injection; Macular Edema; Macular Degeneration; Diabetic Retinopathy; Diabetic Macular Edema
Keywords: Intravitreal Injection; Anesthesia; Macular Degeneration; Diabetic Macular Edema
MeSH Terms: conditions — Macular Edema; Macular Degeneration; Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: A long term safety, dose escalation study design of differing temperatures and duration to test safety and efficacy of cooling anesthesia for intravitreal injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- -15 degrees Celsius for 10 seconds (Experimental): Cooling anesthesia device applied to the eye at -15 degrees Celsius for 10 seconds.
  Interventions: Device: Recens Cooling Anesthesia Device
- -15 degrees Celsius for 15 seconds (Experimental): Cooling anesthesia device applied to the eye at -15 degrees Celsius for 15 seconds.
  Interventions: Device: Recens Cooling Anesthesia Device

INTERVENTIONS:
Device: Recens Cooling Anesthesia Device — Application of cooling anesthesia device prior to intravitreal injection

SUMMARY:
The purpose of this clinical study is to evaluate the long term safety and efficacy of cooling anesthesia application to the eye as anesthesia for intravitreal injection using a novel cooling anesthesia device.

DETAILED DESCRIPTION:
Intravitreal injections have become the standard of care for administering medications for retinal diseases such as age related macular degeneration and diabetic macular edema.

There is considerable apprehension among patients receiving these injections, primarily revolving around adequate anesthesia during the injection. Current methods of anesthesia involve topical anesthetic drops, lidocaine gels, or subconjunctival injections of lidocaine, which suffer from either poor anesthetic effect, corneal irritation, or subconjunctival hemorrhage, as well as significant time for the onset of anesthesia.

Recens Medical has developed a novel medical device which can precisely and rapidly cool the surface of the eye This device cools to a temperature around -5 to -15 degrees Celsius, about the temperature of a cold ice cube, and thus has an excellent safety profile compared to conventional ophthalmic cryotherapy units. The value of such a device is both improved patient comfort, as well as increased efficiency and workflow for retina specialists administering intravitreal injections.

This device has been extensively tested in animal safety studies as well as pilot human studies and has not demonstrated any serious adverse effects and has shown anesthetic effects comparable to current standard of care.

The purpose of this clinical study is to evaluate the long term safety and efficacy of cooling anesthesia application to the eye as anesthesia for intravitreal injection using a novel cooling anesthesia device.

ELIGIBILITY:
Inclusion Criteria:

* Men and women > 18 years old at screening visit.
* Men and women who are undergoing intravitreal injections in either one eye or both eyes with either Lucentis or Eylea as part of their normal standard of care with a 30 gauge needle.
* Subject has received a minimum of 3 intravitreal injections in the study eye prior to the study visit.
* Subject is willing and able to sign the study written informed consent form (ICF).

Exclusion Criteria:

* History of presence of scleromalacia
* Preexisting conjunctival, episcleral or scleral defects
* Less than 18 years of age
* Unable to provide informed consent
* Has received less than 3 injections in the study eye
* Active severe eye disease not controlled with artificial tears and requiring Restasis or other prescription drugs for dry eye.
* History of Endophthalmitis with intravitreal injection
* History of uveitis
* History of retinal detachment in either eye
* History of vitrectomy
* Subjects who received administration of cooling anesthesia as part of the COOL-1 study will not be excluded and are eligible to participate in this study.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Pain of Intravitreal Injection: VAS | Immediately after injection
  Pain of intravitreal injection as measured by 10-point visual analog scale (VAS) (0 meaning no pain, 10 meaning the most severe pain).
Incidence of Anesthesia-Related Adverse Events | 30 minutes after injection
  % of patients that experience cooling anesthesia device-related adverse events, as assessed by anterior segment and posterior segment examination.

SECONDARY OUTCOMES:
Patient Movement During Intravitreal Injection | During injection
  Physician's evaluation of the subject's movement during the intravitreal injection procedure in response to needle penetration (0 = no movement, 1 = mild movement, 2 = marked movement).
Time | Time for entire intravitreal injection procedure
  Recording of the time it takes to perform intravitreal injection procedure.
Patient Anesthetic Preference | 24-48 hours after injection
  Patient response to a questionnaire asking which method of anesthesia they prefer: standard of care or the cooling anesthesia device.
Pain of Intravitreal Injection (Follow-Up): VAS | 24-48 hours after injection
  Pain of intravitreal injection as measured by 10-point visual analog scale (0 meaning no pain, 10 meaning the most severe pain) during follow-up phone call.

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Khanani, MD, Principal Investigator — Sierra Eye Associates
Locations (2):
- United States (2):
  - Sierra Eye Associates, Reno, Nevada
  - Retina Consultants of Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Results of this study will be presented at a national meeting